CLINICAL TRIAL: NCT07104942
Title: Effect of Expiratory Muscle Strength on Hospital Admission, Disease Severity and Quality of Life in Patients With Bronchiectasis
Brief Title: Effect of Expiratory Muscle Strength in Patients With Bronchiectasis
Status: Recruiting | Type: Observational
Sponsor: Nisanur Tutuş (Other)
Responsible Party: Sponsor-Investigator, Nisanur Tutuş, Principal Investigator, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Other Study IDs: bronchiectasis_expiratory
Record Dates: First submitted 2025-07-22; First posted 2025-08-05 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Expiratory muscle strength
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the relationship between expiratory muscle strength and clinical outcomes such as disease severity, hospital admissions, and quality of life in individuals with bronchiectasis.

DETAILED DESCRIPTION:
This study aims to examine the relationship between expiratory muscle strength and clinical outcomes such as disease severity, hospital admission history, and quality of life in individuals with bronchiectasis. Effective coughing is a critical physiological reflex for airway clearance; however, the relationship between expiratory muscle strength and cough effectiveness in the bronchiectasis population has not been clearly established. Identifying expiratory muscle weakness as a potential contributor to increased symptom burden and impaired airway clearance may improve clinical understanding and support the development of targeted physiotherapy interventions. The findings of this study could serve as a foundation for future interventional research in pulmonary rehabilitation and respiratory muscle training for this population.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of non-cystic fibrosis bronchiectasis
* Without an acute infection at the time of assessment (confirmed by medical history, serum C-reactive protein levels, chest X-ray and/or HRCT).
* Being between 18 and 65 years of age

Exclusion Criteria:

* Myopathies
* Stroke (Cerebrovascular accident - CVA)
* Pregnancy
* Unstable cardiac disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Süreyyapaşa Chest Diseases and Chest Surgery Training and Research Hospital
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength | Baseline
  Respiratory muscle function will be assessed by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) in the sitting position using a mouth pressure device (MEC PFT Systems Pocket-Spiro).

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnea Score | Baseline
  Modified Medical Council Dyspnea score will rate the sensation of dyspnea as the person perceives it.The severity of dyspnea is rated on a scale of 0 to 4."0 point" means no dyspnea perception and "4 point" means severe dyspnea perception.
Leicester Cough Questionnaire | Baseline
  This is a short questionnaire that assesses quality of life, particularly for chronic cough. It is relatively easy to administer. The Leicester Cough Questionnaire consists of nineteen questions assessing three different areas: physical, social, and psychological. Scores for the LCQ include mean scores for each domain (ranging from 1 to 7) and a total score calculated as the sum of the domain scores (ranging from 3 to 21). Higher scores indicate better quality of life.
Bronchiectasis Severity Index | Baseline
  The Bronchiectasis Severity Index (BSI) will be used to determine disease severity. This index examines nine parameters: age, body mass index, % predicted FEV1, hospitalizations due to exacerbations in the last 2 years, number of exacerbations in the previous year, level of dyspnea, colonization by Pseudomaonas and other microorganisms, and radiological findings. These scores classify patients into mild (0-4 points), moderate (5-8 points), and severe (9 points and above) groups and identify patients at risk of death, hospitalization and exacerbations.
Hospital Anxiety Depression Scale | Baseline
  This is a 14-item scale developed by Zigmond and Snaith. Seven of these items assess anxiety symptoms, and seven assess depression symptoms. The items in the scale are assessed using a 4-point Likert scale and are based on a scoring system ranging from 0 to 3. Scores range from 0 to 21 for each subscale and can be summed to yield a total anxiety-depression score of up to 42. Higher scores indicate increased symptom severity, while a cut-off score of 8 indicates high levels of depression and anxiety symptoms.
Fatigue severity scale | Baseline
  Individuals' fatigue levels will be assessed using the Fatigue Severity Scale (FSS). The FSS consists of 9 questions scored on a 7-point Likert scale, indicating a perceived level of fatigue that may require medical attention. It is a valid and reliable instrument, with a score of 7 being associated with greater fatigue.
Spirometric measurements (Forced vital capacity) | Baseline
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. Forced vital capacity (FVC): the maximum amount of air that can be forcibly exhaled from the lungs after fully inhaling. It can be recorded in percentages or liters.
Spirometric measurements (First second forced expiratory volume) | Baseline
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. First-second forced expiratory volume (FEV1): the amount of air that can be exhaled with force in 1 second. It can be recorded in percentages or liters.
Spirometric measurements (FEV1/FVC ratio) | Baseline
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. It is calculated by dividing FEV1 by FVC. It is expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Süreyyapaşa Chest Diseases and Chest Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided